CLINICAL TRIAL: NCT01022606
Title: Intra-arterial Measurement of pO2 in Walking Induced Transient Hack ("WITH") Profiles
Brief Title: Intra-arterial Measurement of pO2 in Walking Induced Transient Hack Profiles
Acronym: Initial-VHS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Stopped for one complication event (arterial occlusion)
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: PE 2009-16
Record Dates: First submitted 2009-11-24; First posted 2009-12-01 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Claudication
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with walking limitation (Other): Patients with claudication and Walking-Induced Transient Hack (W.I.T.H.) tcpO2 profiles are tested on treadmill with invasive pO2 arterial sampling and body temperature recording
  Interventions: Other: Arterial sampling

INTERVENTIONS:
Other: Arterial sampling — Arterial pO2 (ABL5) Body Temperature (Vitalsens Cortemp) tcpO2 TCM400
  Other Names: All material is CE marked and approved for huamn use

SUMMARY:
Confirm with invasive measurement the presence of a Walking-Induced Transient Hack (WITH) profile

DETAILED DESCRIPTION:
Arterial PO2 and body temperature measurements during exercise

ELIGIBILITY:
Inclusion Criteria:

* walking induced transient Hack (WITH) tcpO2 profile

Exclusion Criteria:

* rejection by patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
arterial pO2 | 2 months (time required to organise the test)

CONTACTS AND LOCATIONS:
Overall Officials: P Abraham, MD, PhD, Study Chair — University Hospital
Locations (1):
- University Hospital, Angers, France